CLINICAL TRIAL: NCT05700370
Title: Equivalency of MyProstateScore (MPS) Results Between Urine Samples Collected With or Without a Preceding Digital Rectal Examination
Brief Title: MyProstateScore Equivalency With and Without DRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: LynxDx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Equivalency-Study-001
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: biomarker; tumor; prostate; prostatic neoplasm; prostate-specific antigen; early detection of cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sample collected with preceding DRE, then without (Experimental): All subjects participate in the control and experimental collection event sequentially. The control group will consist of urine samples collected post-DRE, and the experimental group will consist of urine samples collected by the same subjects without preceding DRE.
  Interventions: Diagnostic Test: MyProstateScore

INTERVENTIONS:
Diagnostic Test: MyProstateScore — MyProstateScore is a urine-based biomarker test used to predict the risk of clinically significant prostate cancer

SUMMARY:
The purpose of the study is to quantify the concordance of MPS results between first-catch urine samples collected post-DRE and those collected without a DRE.

DETAILED DESCRIPTION:
The process for obtaining a urine sample for MPS currently requires a DRE within one hour prior to urine collection. We aim to understand whether a DRE is a required step prior to urine collection for MPS, and to explore alternative methods that may eliminate the need for a DRE. In order to do so, we will perform a crossover study in which each subject provides a sample under both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for prostate biopsy (Bx)
* If Bx naïve and ≤75yo then PSA 3-10 ng/mL
* If Bx naïve and >75yo then PSA 4-10 ng/mL
* If prior negative Bx then PSA may exceed 10 ng/mL
* If DRE very suspicious, then PSA below the thresholds of 3 ng/mL (≤75yo) and 4 ng/mL (>75yo) are acceptable

Exclusion Criteria:

- Prior diagnosis of prostate cancer

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
MPS equivalency with and without DRE | Study participation will span 8 days
  The process for obtaining a urine sample for MPS currently requires a DRE within one hour prior to urine collection. We aim to understand whether a DRE is a required step prior to urine collection for MPS, and to explore alternative methods that may eliminate the need for a DRE.
MPS validity rate with and without DRE | Study participation will span 8 days
  Rate of invalid test result equivalency in post-DRE versus non-DRE paired urine samples. Rate will be measured as the percentage of subjects who return an invalid urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Patel, MD, Principal Investigator — Arizona State Urological Institute
Locations (1):
- Arizona State Urological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
MPS results from the post-DRE urine sample will be reported to the provider, consistent with current commercially available processes. Results from the experimental sample collected without a preceding DRE will not be reported to the subject or their provider.
Time Frame: In accordance with the commercially available process
Access Criteria: In accordance with the commercially available process